CLINICAL TRIAL: NCT01158248
Title: A Two-Stage Multicenter Phase II Trial of Concurrent Panitumumab Immunotherapy, Cisplatin Chemotherapy and Pelvic Radiotherapy for Primary Cancer of the Uterine Cervix Stage IB-IIIB
Brief Title: Panitumumab, Cisplatin, and Pelvic Radiation Therapy in Treating Patients With Stage IB, Stage II, or Stage III Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000675699; MUI-AGO-20; EUDRACT-2009-012453-38; EU-21043
Record Dates: First submitted 2010-07-07; First posted 2010-07-08 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-07

CONDITIONS: Cervical Cancer
Keywords: cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical small cell carcinoma; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Panitumumab; Cisplatin; Brachytherapy

INTERVENTIONS:
Biological: panitumumab
Drug: cisplatin
Radiation: brachytherapy
Radiation: external beam radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving panitumumab and cisplatin together with pelvic radiation therapy may be effective in treating patients with cervical cancer.

PURPOSE: This phase II trial is studying the side effects of giving panitumumab and cisplatin together with pelvic radiation therapy in treating patients with stage IB, stage II, or stage III cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the activity of concurrent panitumumab and cisplatin chemoradiotherapy in patients with stage IB-IIIB, KRAS-wild type (KRAS^wt) cervical cancer, in terms of progression-free survival at 4 months by MRI according to RECIST criteria.
* To assess the rate of skin toxicity (e.g., photosensitivity, acneiform rash, and dermatitis) CTCAE grade 4 and/or gastrointestinal toxicity (comprising all grades of gastrointestinal perforation; leakage of stomach, small intestine, colon, rectum, or elsewhere in the peritoneal cavity occurring after the first application of study treatment and not immediately related to a surgical procedure) at 4 months, of this regimen in these patients.

Secondary

* To assess the activity of this regimen in KRAS^wt-positive and -negative patients, in terms of overall response rate at 4 months.
* To assess the activity of this regimen in KRAS^wt-positive and -negative patients, in terms of progression-free survival at 12 months and 24 months.
* To assess the activity of this regimen in KRAS^wt-positive and -negative patients, in terms of overall survival at 12 months and 24 months.
* To assess the rate of severe adverse events of this regimen in patients with KRAS^wt and KRAS-mutant gene status at 4 months.
* To assess the rate of post-treatment severe adverse events at 12 months and 24 months.
* To assess the rate of severe adverse events of panitumumab monotherapy at day 14.

OUTLINE: This is a multicenter study.

Patients receive panitumumab IV on days 1, 14, 29, and 43 and cisplatin IV on days 14, 22, 29, 36, 43, and 50 in the absence of disease progression or unacceptable toxicity. Patients undergo concurrent external-beam and intracavitary radiotherapy (teletherapy of pelvis or high-dose rate brachytherapy) according to treating center specific standards.

Blood and tissue specimens are collected periodically for laboratory analysis.

After completion of study treatment, patients are followed periodically for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed cervical cancer, including the following subtypes:

  * Squamous small-cell or large-cell carcinoma
  * Adenosquamous cell carcinoma
  * Adenocarcinoma
  * Keratinizing or non-keratinizing carcinoma
* Stage IB-IIIB disease
* No para-aortic lymph node metastases or clinical indication for para-aortic field irradiation
* No predominant and clinically effective neuroendocrine tumor cell differentiation

PATIENT CHARACTERISTICS:

* WH0 performance status 0-2
* Serum creatinine clearance > 50 mL/min
* No other prior or current malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or carcinoma in-situ of the cervix
* No acute life-threatening vaginal hemorrhage (requiring emergency irradiation or RBC transfusion)

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 4 months by MRI according to RECIST criteria
Rate of skin and/or gastrointestinal toxicity CTCAE grade 4 at 4 months

SECONDARY OUTCOMES:
Overall response rate at 4 months according to RECIST criteria
Progression-free survival at 12 and 24 months according to RECIST criteria
Overall survival at 12 and 24 months
Rate of severe adverse events according to CTCAE at 4 months
Rate of post-treatment severe adverse events according to CTCAE at 12 and 24 months
Rate of severe adverse events according to CTCAE of panitumumab monotherapy at day 14

CONTACTS AND LOCATIONS:
Overall Officials: Alain Zeimet, Principal Investigator — Medical University Innsbruck
Locations (1):
- Innsbruck Universitaetsklinik, Innsbruck, Austria